CLINICAL TRIAL: NCT02696720
Title: A Randomized Controlled Trial of Lidocaine Patch for Lower Limb Amputation Pain
Brief Title: A Trial of Lidocaine Patch for Lower Limb Amputation Pain
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Samar Hatem, Head of clinic, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHUB-patch lidocaine
Record Dates: First submitted 2016-02-26; First posted 2016-03-02 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Phantom Limb Pain (PLP); Primary/Secondary Scar Hyperalgesia
Keywords: lidocaine; phantom limb pain (PLP); Primary/secondary scar hyperalgesia
MeSH Terms: conditions — Phantom Limb | interventions — Lidocaine; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine (Experimental): During a period of six weeks, a lidocaine patch will be applied around the wound (cut in two parts, 1cm above and below the wound, without direct contact with the scar) for a total of twelve hours per day, during night time.
  Interventions: Drug: Lidocaine
- Sham (Sham Comparator): During a period of six weeks, a visually identical patch (sham) will be applied around the wound (cut in two parts, 1cm above and below the wound, without direct contact with the scar) for a total of twelve hours per day, during night time.
  Interventions: Other: Sham

INTERVENTIONS:
Drug: Lidocaine
  Arms: Lidocaine
Other: Sham
  Arms: Sham

SUMMARY:
Phantom limb pain (PLP) and scar hyperalgesia (SH) are frequent problems after amputation; in particular most persons who undergo limb amputation will experience phantom pain. The neuropathic nature of PLP suggests the involvement of both peripheral and central neurological mechanisms, including neuroplastic changes in the central nervous system. PLP as other central nervous system-related pain syndromes remains a challenge for treatment. Scar hyperalgesia involves peripheral mechanisms and results frim the production of substances liberated by damaged skin cells. These inflammatory substances lower the pain threshold by altering the chemical environment of skin nerve endings. Scan hyperalgesia is associated with secondary mechanical hyperalgesia in the skin area around the scar.

The lidocaine patch 5% is a topical analgesic acting by blocking sodium channels of peripheral nerve endings and by inhibiting ectopic discharges in sensitized and hyperactive cutaneous nociceptors. The patch is noninvasive, with minimal systemic absorption resulting in a reduced risk of drug-drug interaction. In addition, a central analgesic effect of lidocaine has been suggested. The lidocaine patch 5% is currently licensed for the treatment of symptomatic postherpetic neuralgia. It also has been successfully used in patients with other neuropathic pain states, such as entrapment neuropathies, painful idiopathic distal sensory polyneuropathies and postoperative/post traumatic neuropathic chronic cutaneous pain. The lidocaine patch has not been studied for the management and prevention of phantom limb pain.

The aim of the present research is to investigate if a lidocaine patch 5% is effective for reducing PLP and primary/secondary scar hyperalgesia. The hypothesis is that persistent peripheral nociceptive input from the stump after surgery may drive maladaptive cortical reorganization leading to chronic central pain and thus promote chronic phantom limb pain. Treating scar hyperalgesia on the stump with topical lidocaine may reduce the activity of peripheral nociceptive afferents and thus decrease the likelihood of developing persistent phantom limb pain.

This study is designed as a randomized controlled multicentric double blind trial, in which the effectiveness of applying a 5% lidocaine patch for 6 weeks will be compared with a sham.

ELIGIBILITY:
Inclusion Criteria:

* All above or below knee amputations , two months or more after surgery, after complete wound healing (no clips, no stitches, no seepage)

Exclusion Criteria:

* History of central nervous system disease
* History of major psychiatric disease (MMS<23/30, HADS>8/21)
* Pregnancy
* Known hypersensitivity to local anesthetics (lidocaine, bupivacaine, etidocaine, mepivacaine, prilocaine)
* skin irritation on the stump

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05-13 (Actual); Primary Completion 2017-06-13 (Actual); Study Completion 2017-06-13 (Actual)

PRIMARY OUTCOMES:
Patient-reported overall daily pain intensity | Daily, starting seven days before patch placement (baseline) till six weeks after patch placement
  The overall daily pain intensity (stump, scar and phantom pain combined) will be rated on a 0 to 100 visual analogue scale with anchors of 0 (no pain) to 100 (worst pain ever experienced).

SECONDARY OUTCOMES:
Neuropathic Pain (DN4) | at baseline - 7 days before patch placement
  Screening for neuropathic pain, by using the DN4 questionnaire
Neuropathic pain | at baseline - 7 days before patch placement
  Rated with the Neuropathic Pain Symptom Inventory
Neuropathic pain | One day after patch placement
  Rated with the Neuropathic Pain Symptom Inventory
Neuropathic pain | 6 weeks after patch placement
  Rated with the Neuropathic Pain Symptom Inventory
Neuropathic pain | 6 months after patch placement
  Rated with the Neuropathic Pain Symptom Inventory
Pain (McGill) | at baseline - 7 days before patch placement
  Rated by the Short-Form McGill Pain Questionnaire, sensitive to the effects of pain treatment.
Pain (McGill) | One day after patch placement
  Rated by the Short-Form McGill Pain Questionnaire, sensitive to the effects of pain treatment.
Pain (McGill) | 6 weeks after patch placement
  Rated by the Short-Form McGill Pain Questionnaire, sensitive to the effects of pain treatment.
Quality of life | at baseline -7 days before patch placement
  Rated by the SF36 questionnaire
Quality of life | six weeks after patch placement
  Will be rated by the SF36 questionnaire
Quality of life | six months after patch placement
  Will be rated by the SF36 questionnaire
Sleep quality | baseline -7 days before patch placement
  will be assessed with the Pittsburgh Sleep Quality index
Sleep quality | 6 weeks after patch placement
  will be assessed with the Pittsburgh Sleep Quality index
Sleep quality | 6 months after patch placement
  will be assessed with the Pittsburgh Sleep Quality index
Delay of dress of provisory prosthesis | From the day of the surgery till the day of the delivery of temporary prosthesis, for a maximum of 6 months
  Number of days between surgery and delivery of temporary prosthesis
Delay of dress of provisory prosthesis | From the day of patient inclusion in the research protocol till the day of the delivery of temporary prosthesis, for a maximum of 6 months
  Number of days between inclusion in the research protocol and delivery of temporary prosthesis
Cumulative analgesic consumption (morphine equivalents) | baseline -7 days before patch placement
  Rated by the cumulative analgesic consumption score (CACS)
Cumulative analgesic consumption (morphine equivalents) | 1 day after patch placement
  Rated by the cumulative analgesic consumption score (CACS)
Cumulative analgesic consumption (morphine equivalents) | 6 weeks after patch placement
  Rated by the cumulative analgesic consumption score (CACS)
Phantom Limb Pain occurence | 6 months after patch placement
  occurence of phantom limb pain

CONTACTS AND LOCATIONS:
Overall Officials: Samar Hatem, MD, Principal Investigator — CHU Brugmann; Simone Brienza, MD, Principal Investigator — CHU Brugmann; Valérie Gangji, MD, Principal Investigator — Erasme
Locations (2):
- Belgium (2):
  - CHU Brugmann - Queen Astrid, Brussels
  - Erasme -CTR, Brussels

REFERENCES:
- [Background] Robinson LR, Czerniecki JM, Ehde DM, Edwards WT, Judish DA, Goldberg ML, Campbell KM, Smith DG, Jensen MP. Trial of amitriptyline for relief of pain in amputees: results of a randomized controlled study. Arch Phys Med Rehabil. 2004 Jan;85(1):1-6. doi: 10.1016/s0003-9993(03)00476-3. PMID 14970960
- [Background] HARDY JD, WOLFF HG, GOODELL H. Experimental evidence on the nature of cutaneous hyperalgesia. J Clin Invest. 1950 Jan;29(1):115-40. doi: 10.1172/JCI102227. No abstract available. PMID 15399521
- [Background] Gammaitoni AR, Alvarez NA, Galer BS. Safety and tolerability of the lidocaine patch 5%, a targeted peripheral analgesic: a review of the literature. J Clin Pharmacol. 2003 Feb;43(2):111-7. doi: 10.1177/0091270002239817. PMID 12616661
- [Background] Koppert W, Ostermeier N, Sittl R, Weidner C, Schmelz M. Low-dose lidocaine reduces secondary hyperalgesia by a central mode of action. Pain. 2000 Mar;85(1-2):217-24. doi: 10.1016/s0304-3959(99)00268-7. PMID 10692621
- [Background] Nalamachu S, Crockett RS, Gammaitoni AR, Gould EM. A comparison of the lidocaine patch 5% vs naproxen 500 mg twice daily for the relief of pain associated with carpal tunnel syndrome: a 6-week, randomized, parallel-group study. MedGenMed. 2006 Aug 9;8(3):33. PMID 17406167
- [Background] Herrmann DN, Barbano RL, Hart-Gouleau S, Pennella-Vaughan J, Dworkin RH. An open-label study of the lidocaine patch 5% in painful idiopathic sensory polyneuropathy. Pain Med. 2005 Sep-Oct;6(5):379-84. doi: 10.1111/j.1526-4637.2005.00058.x. PMID 16266359
- [Background] Hans G, Joukes E, Verhulst J, Vercauteren M. Management of neuropathic pain after surgical and non-surgical trauma with lidocaine 5% patches: study of 40 consecutive cases. Curr Med Res Opin. 2009 Nov;25(11):2737-43. doi: 10.1185/03007990903282297. PMID 19788351
- [Background] Bouhassira D, Attal N, Alchaar H, Boureau F, Brochet B, Bruxelle J, Cunin G, Fermanian J, Ginies P, Grun-Overdyking A, Jafari-Schluep H, Lanteri-Minet M, Laurent B, Mick G, Serrie A, Valade D, Vicaut E. Comparison of pain syndromes associated with nervous or somatic lesions and development of a new neuropathic pain diagnostic questionnaire (DN4). Pain. 2005 Mar;114(1-2):29-36. doi: 10.1016/j.pain.2004.12.010. Epub 2005 Jan 26. PMID 15733628
- [Background] Bouhassira D, Attal N, Fermanian J, Alchaar H, Gautron M, Masquelier E, Rostaing S, Lanteri-Minet M, Collin E, Grisart J, Boureau F. Development and validation of the Neuropathic Pain Symptom Inventory. Pain. 2004 Apr;108(3):248-257. doi: 10.1016/j.pain.2003.12.024. PMID 15030944
- [Background] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771